CLINICAL TRIAL: NCT01627990
Title: The Compatibility of Nivestim™ Under Cytotoxic Chemotherapy in the Treatment of Malignant Diseases
Brief Title: Nivestim™ in Treatment of Malignant Diseases
Status: Completed | Type: Observational
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: VENICE
Record Dates: First submitted 2012-06-07; First posted 2012-06-26 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Solid Tumour; Malignant Haematological Tumour; Primary or Secondary Prophylactic Treatment
Keywords: cytotoxic chemotherapy; G-CSF; Solid tumour; Malignant haematological tumour

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * CD34+ cell count in peripheral blood (low/high at Visit 1)
  * Concentrations of haemoglobin, thrombocytes, leukocytes, neutrophil and CRP are represented across time (v1, 2 and 3)
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to observe the tolerability, safety and efficacy of preventative treatment using Nivestim™ in patients receiving cytotoxic chemotherapy for cancer.

DETAILED DESCRIPTION:
This is a non-interventional, descriptive, national, multi-site, longitudinal and prospective observational study with in-patients adults or minors undergoing cytotoxic chemotherapy, being treated prophylactically with Nivestim™ in order to reduce the duration of neutropenia and to reduce the incidence of chemotherapy-induced Febrile neutropenia (FN).

ELIGIBILITY:
Inclusion Criteria:

* No age limit
* Declaration of informed consent signed by patient or legal guardian
* Patients with a solid tumour or with a malignant haematological tumour
* Patients for whom cytotoxic chemotherapy is planned, irrespective of cycle
* Patients who are due to undergo, or who should undergo, (primary or secondary) prophylactic treatment using Nivestim™, either to shorten the duration of a neutropenia or to prevent the occurrence of chemotherapy induced febrile neutropenia (FN).

Exclusion Criteria:

* Patients with chronic myeloid leukaemia (CML) or with myelodysplastic Syndrome (MDS)
* Patients who are hypersensitive to the active substance or to one of the excipients of Nivestim™
* Patients not undergoing chemotherapy
* Patients being treated curatively with Granulocyte-Colony Stimulating Factor (G-CSF)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children and adult patients with a solid tumour or a malignant haematological tumour
Sampling Method: Non-Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Incidence of hospitalisation due to febrile neutropenia and/or infection | 6 months

SECONDARY OUTCOMES:
Characterisation of patients being treated with Nivestim™ | 6 months
  Characterisation of patient based on:
  * Socio-demographic data
  * previous medical history (Surgical and therapeutic)
  * Tumour data
  * Chemotherapy data
  * Clinical and laboratory data preceding treatment with Nivestim™
Treatment with Nivestim™ as part of daily routine | 6 months
  * Therapeutic indication
  * Dosage and mode of administration
  * Duration of treatment (planned and carried through)
  * Delay in start of treatment since last chemotherapy for purposes of prophylaxis
  * Absolute Neutrophil Count (ANC) during study.
Description of the efficacy of treatment with Nivestim™ | 6 months
  Description of the efficacy of treatment with Nivestim(TM) which includes the following parameters:
  * Duration of neutropenia
  * Incidence of febrile neutropenia
  * Frequency of infection
  * Delay in chemotherapy cycles due to neutropenia
  * Reduction in chemotherapy doses due to neutropenia
  * Assessment of patient
Detailed description of tolerability and safety | 6 months
  * Hospitalisation
  * Adverse events
Description of the characteristics of the participating physicians | During the study initiation visit
  Socio-demographic data (age, gender, field of specialisation, structure of practice, title)
Prescription routine of G-CSF (Granulocyte Colony-Stimulating Factor) | During the study initiation visit
  Criteria for selecting Nivestim™

CONTACTS AND LOCATIONS:
Locations (48):
- Germany (48):
  - Facharzt für Innere Medizin, Onkologie, Hämatologie, Ahaus
  - Studienzentrum Hämatologie/Onkologie/Diabetologie, Aschaffenburg
  - Facharzt für Innere Medizin Hämatologie / Onkologie, Bad Säckingen
  - MediOnko-Institut GbR, Berlin
  - Onkoplan GmbH/Onkologische Schwerpunkpraxis, Berlin
  - FA f. Frauenheilkunde und Geburtshilfe Gynäkologische Onkologie, Chemnitz
  - MVZ Delitzsch GmbH, Delitzsch
  - Gesellschaft für onkologische Studien Dortmund mbH, Dortmund
  - Gemeinschaftspraxis, Dresden
  - Gemeinschaftspraxis Haematologie/Medizin Onkologie, Düsseldorf
  - Gemeinschaftspraxis, Eisenach
  - Krankenhaus Nordwest GmbH Institut für klinische Forschung, Frankfurt am Main
  - Internist - Hämatologe - Onkologe, Garbsen
  - Onkodok GmbH, Gütersloh
  - Fachärztin für Allgemeinmedizin, Hamburg
  - Facharzt für innere Medizin, Hamburg
  - Internist - Hämatologe - Onkologe, Hanover
  - ODZ-Petersen GmbH, Heidenheim
  - DOKUSAN Gesellschaft für medizinische Studien mbH & Co. KG, Herne
  - ZAGO, Krefeld
  - FA f. Frauenheilkunde und Geburtshilfe, Leipzig
  - Pneumologisch/onkologisch/internistisches Studienzentrum, Leipzig
  - Fachübergreifende Gemeinschaftspraxis Innere Medizin, Hämatologie, Onkologie, Tumortherapie, Palliativmedizin, Lippstadt
  - Praxis für Innere Medizin, Hämatologie und Onkologie, Mainz
  - Johannes Esling Klinikum Minden, Minden
  - OnkoLog Moers GbR, Moers
  - Fachärzte für Innere Medizin - Hämatologie u. Internistische Onkologie - Bluttransfusionswesen, München
  - Forschungs- und Studiengesellschaft HOPE München GmbH, München
  - Münster
  - FÄ für Innere Medizin Hämatologie/Internistische Onkologie, Neustadt A. Rbge
  - Facharzt für Innere Medizin - Medikamentöse Tumortherapie - Palliativmedizin, Neustadt/Sachsen
  - MVZ Nordhausen gGmbH/ FA für Frauenheilkunde und Geburtshilfe, Nordhausen
  - Martha-Maria Krankenhaus gGmbH MVZ Onkologie, Nuremberg
  - Fachärztin für Innere Medizin Hämatologie u. Internistische Onkologie, Oelde
  - Onkologische Praxis Oldenburg/ Delmenhorst, Oldenburg
  - Medizinisches Versorgungszentrum Onkologische Schwerpunktpraxis, Olpe
  - Osnabrück
  - Facharzt für Innere Medizin - Hämatologie - Onkologie - Medikamentöse Tumortherapie, Remscheid
  - Frauenärzte -Naturheilverfahren-, Rodgau
  - Facharzt für Fraueneheilkunde und Geburtshilfe Gynäkologische Onkologie, Scheibenberg
  - Onkol. Managementgesellschaft Bonn/Rhein-Sieg/Ahr mbH, Siegburg
  - Medizinisches Versorgungszentrum GbR, Soest-Paradiese
  - g.SUND Gyn. Kompetenzzentrum FA f. Frauenheilkunde & Geburtshilfe SP Gynäkologie Onkologie operative Gyn./ med. Tumortherapie/ Palliativmed., Stralsund
  - Stuttgart
  - Fachärzte für Innere Medizin -Hämatologie und Internistische Onkologie, Velbert
  - Gesellschaft zur Förderung von Wissenschaft und Qualitätssicherung in der ambulanten Onkologie (GFWQ), Wiesbaden
  - FA f. Frauenheilkunde u. Geburtshilfe Marien-Hospital Witten gGmbH, Witten
  - FA für innere Medizin/Hämatologie und Int. Onkologie/Palliativmedizin, Zittau

REFERENCES:
- [Derived] Fruehauf S, Otremba B, Stotzer O, Rudolph C. Compatibility of Biosimilar Filgrastim with Cytotoxic Chemotherapy during the Treatment of Malignant Diseases (VENICE): A Prospective, Multicenter, Non-Interventional, Longitudinal Study. Adv Ther. 2016 Nov;33(11):1983-2000. doi: 10.1007/s12325-016-0419-1. Epub 2016 Oct 14. PMID 27743353
- [Derived] Kamioner D, Fruehauf S, Maloisel F, Cals L, Lepretre S, Berthou C. Study design: two long-term observational studies of the biosimilar filgrastim Nivestim (Hospira filgrastim) in the treatment and prevention of chemotherapy-induced neutropenia. BMC Cancer. 2013 Nov 16;13:547. doi: 10.1186/1471-2407-13-547. PMID 24237790